CLINICAL TRIAL: NCT04982718
Title: Randomized Controlled Trial of Home-based Hepatitis C Self-testing for Key Populations in Malaysia
Brief Title: HCV Self-testing in Malaysia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Hospital Sultanah Bahiyah (Other Government); Ministry of Health, Malaysia (Other Government); Malaysian AIDS Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: HC021
Record Dates: First submitted 2021-07-16; First posted 2021-07-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C; Diagnostic Self Evaluation
Keywords: Linkage to care; Online self-test distribution; Self-test
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention or control group in a 2:1 ratio. In the intervention group, participants will receive a HCV self-test (ST) kit delivered in non-identifiable packaging to their home or a preferred mailing address. In order to evaluate two sampling methods for HCV self-testing, the first 250 participants in the intervention group will receive an oral fluid-based HCV ST, and the next 250 participants will receive a blood-based fingerstick HCV ST. In the control group, participants will receive information about standard of care HCV antibody testing available at local testing sites in their community and information about additional supporting materials, such as access to live chat and a call center for questions about testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral fluid-based HCV ST (Experimental): In the intervention group, participants will receive a HCV self-test (ST) kit delivered in non-identifiable packaging to their home or a preferred mailing address. The kit will include the test, instructions for use, and information about additional supporting materials, such as access to live chat and a call center for questions about testing. In order to evaluate two sampling methods for HCV self-testing, the first 250 participants in the intervention group will receive an oral fluid-based HCV ST.
  Interventions: Diagnostic Test: OraQuick® HCV Self-Test
- Blood-based HCV ST (Experimental): In the intervention group, participants will receive a HCV self-test (ST) kit delivered in non-identifiable packaging to their home or a preferred mailing address. The kit will include the test, instructions for use, and information about additional supporting materials, such as access to live chat and a call center for questions about testing. In order to evaluate two sampling methods for HCV self-testing, the next 250 participants will receive a blood-based fingerstick HCV ST.
  Interventions: Diagnostic Test: First Response® HCV Self-Test
- Control standard of care (No Intervention): In the control group, participants will receive information about standard of care HCV antibody testing available at local testing sites in their community and information about additional supporting materials, such as access to live chat and a call center for questions about testing.

INTERVENTIONS:
Diagnostic Test: OraQuick® HCV Self-Test — Self-testing will be performed using the OraQuick® HCV Self-Test manufactured by OraSure Technologies Inc., USA. Modified IFU developed by the manufacturer will be used to adapt the below professional use kits to a self-test: the OraQuick® HCV Rapid Antibody Test is prequalified by WHO and CE marked for professional use (sensitivity 98.1%, specificity 99.6%).
  As it is not approved for self-test use in Malaysia, the OraQuick® HCV Self-Test kits provided to participants in the intervention group will be labelled for Research Use Only (RUO) and test results will not be used for patient management.
  Arms: Oral fluid-based HCV ST
Diagnostic Test: First Response® HCV Self-Test — Self-testing will be performed using the First Response® HCV Card Test (Self Test) manufactured by Premier Medical Corporation, India. Modified IFU developed by the manufacturer will be used to adapt the below professional use kits to a self-test: the First Response® HCV Card Test is CE-marked and currently under WHO review for professional use (sensitivity 100%, specificity 100%).
  As it is not approved for self-test use in Malaysia, the First Response® HCV Self-Test kits provided to participants in the intervention group will be labelled for Research Use Only (RUO) and test results will not be used for patient management.
  Arms: Blood-based HCV ST

SUMMARY:
Self-testing with easy-to-use rapid diagnostic tests (RDTs) has been successfully used for diseases such as HIV. The availability of self-testing has been shown to increase testing rates and testing acceptability in diverse populations around the world, in large part due to its convenience and privacy advantages. Self-testing has also been effectively used to reach key populations who may not be covered by traditional healthcare programs, such as persons who inject drugs and men who have sex with men. In Malaysia, HIV self-testing has been shown to have moderate to high levels of acceptability, depending on the population, test used, and test delivery framework. In the present study we aim to evaluate the acceptability and impact of an online program enabling home-based hepatitis C virus (HCV) self-testing in Malaysia.

DETAILED DESCRIPTION:
Malaysia is an upper middle-income country with a population of more than 32 million, comprising thirteen states and three federal territories. It is estimated that the hepatitis C virus (HCV) seroprevalence in the general population of Malaysia is between 0.3% and 2.5%. In Malaysia, people who inject drugs represent just 0.24% (75 000) of the adult population; however, they are disproportionately affected by HCV, with an overall HCV prevalence of 67.5% to 89.9%. Other key populations in Malaysia at higher risk of HCV include 77 903 people living with human immunodeficiency virus (HIV, 0.24%), 221 698 men who have sex with men (0.69%), 22 000 female sex workers (0.069%), and 15 000 transgender sex workers (0.047%).

The major challenges faced by Malaysia in eliminating viral hepatitis have been under-screening, under-diagnosis and under-treatment. A high proportion of those infected with HCV remain undiagnosed and, until 2018, only a small proportion of those infected received treatment each year. Up until 2017, it is estimated that just 6.1% (23 258) of people infected with HCV were diagnosed.

Self-testing with easy-to-use rapid diagnostic tests (RDTs) has been successfully used for diseases such as HIV. The availability of self-testing has been shown to increase testing rates and testing acceptability in diverse populations around the world, in large part due to its convenience and privacy advantages. In the present study we aim to evaluate the acceptability and impact of an online program enabling home-based HCV self-testing in Malaysia.

FIND, in conjunction with the Malaysian AIDS Council (MAC) and the Ministry of Health (MOH) Malaysia, is evaluating HCV self-testing as a way to expand outreach, improve HCV testing rates, and increase linkage to care among HCV-infected individuals. The ability to utilize an existing online platform promoting HIV self-testing (JomTest) will enable us to examine how offering home-based HCV self-testing may help identify HCV-infected individuals and link them to care. *The online platform JomTest is currently hosting a research study with Medical Research Ethics Committee, University Malaya Medical Center MRECID No. 202013-8135, study title "Integrated HIV self-testing (HIVST) service delivery in Malaysia for policy and service development: JomTest online" and aims to assess the integrated HIVST service delivery in Malaysia for policy and service development through the platform.

This study will evaluate the impact of a home-based HCV self-testing program in Malaysia. We aim to describe the acceptability and impact of an online platform offering home-based HCV self-tests to key populations. Since HCV self-tests detect the presence of antibodies to HCV, indicating exposure to HCV, any individual reporting a positive HCV self-test will be referred to HCV RNA confirmatory testing in order to identify active HCV infection. Those confirmed to have active HCV infection with a positive HCV RNA test will be linked to HCV treatment and care. Rates of testing and linkage to care will be measured, along with knowledge, attitudes, and practices around HCV testing and care.

This is a randomized controlled trial comparing an online platform providing home-delivery of HCV self-tests to referral to standard of care community-based HCV testing sites in Malaysia. Study participants will be recruited through an existing HIV self-testing program using an online platform JomTest. Interested participants will sign up and proceed for study eligibility screening and if eligible, proceed to complete an online consent form. All consented and enrolled study participants will complete an online baseline survey collecting demographics and knowledge and attitudes towards HCV testing.

Participants will be randomized to the intervention or control group in a 2:1 ratio. In the intervention group, participants will receive a HCV self-test (ST) kit delivered in non-identifiable packaging to their home or a preferred mailing address. The kit will include the test, instructions for use, and information about additional supporting materials, such as access to live chat and a call center for questions about testing. In order to evaluate two sampling methods for HCV self-testing, the first 250 participants in the intervention group will receive an oral fluid-based HCV ST, and the next 250 participants will receive a blood-based fingerstick HCV ST. In the control group, participants will receive information about standard of care HCV antibody testing available at local testing sites in their community and information about additional supporting materials, such as access to live chat and a call center for questions about testing.

As there is no quality-assured HCV self-test today, the professional use OraQuick® HCV Rapid Antibody Test and First Response® HCV Card Test that have been repackaged and labelled with Instructions for Use (IFU) adapted by the manufacturers for self-testing would be used in this study. The OraQuick® HCV Rapid Antibody Test is prequalified by WHO and CE marked for professional use (sensitivity 98.1%, specificity 99.6%); the First Response® HCV Card Test is CE-marked and currently under WHO review for professional use (sensitivity 100%, specificity 100%). Both these professional tests are not yet registered with the Medical Device Authority in Malaysia. The OraQuick® HCV Self-Test and First Response® HCV Self-Test kits provided to participants in the intervention group will be labelled for Research Use Only (RUO).

All participants will be sent a reminder for online Follow-up survey #1 and the opportunity to upload any testing result in approximately 2-4 weeks from day of enrolment. A second online Follow-up survey #2 will be sent after the closure of the first survey. Up to 3 reminders may be sent if a survey has not been completed. Participants will receive 20 Ringgit (~5 USD) for completing Follow-up survey #1 and an additional 20 Ringgit for completion of the Follow-up survey #2. Any participants found to be HCV antibody positive through the study will be supported to access HCV management and care services for confirmatory HCV testing and HCV treatment if required and be provided additional assistance through MAC's existing peer navigation system as outlined in the organization's standard operating procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eligible to access services on the JomTest online platform
* Not known to be HCV antibody positive
* Not tested for HCV within the last 6 months
* Able to read and understand Bahasa Malaysia or English
* Able to understand the scope of the study and provide online informed consent

Exclusion Criteria:

• Self-reported previously confirmed positive HCV status (either antibody or RNA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of home-based HCV self-testing on the uptake of HCV antibody testing | Time Frame: 2 weeks to 2 months after enrollment
  The number and estimate of the proportion of participants who report completing the HCV antibody testing in the intervention group vs the control group.
To assess the impact of home-based HCV self-testing on the uptake of HCV antibody testing | Time Frame: 2 weeks to 2 months after enrollment
  To assess that the proportion of participants who report completing the HCV antibody testing in the intervention group is superior to that of the participants in the control group by a margin of 20%.

SECONDARY OUTCOMES:
To assess the impact of HCV self-testing on the number of HCV antibody positive individuals who are aware of their status | 2 weeks to 2 months after enrollment
  Number and estimate of the proportion of HCV antibody positive individuals made aware of their status in the intervention vs control group
To assess the impact of HCV self-testing on linkage and completion of HCV RNA confirmatory testing in HCV antibody positive individuals | 2 weeks to 6 months after enrollment
  Number and estimate of the proportion of HCV antibody positive individuals who are referred to and complete HCV RNA confirmatory testing in the intervention vs control group
To assess the impact of HCV self-testing on treatment initiation in HCV RNA positive individuals eligible to start treatment | 2 weeks to 6 months after enrollment
  Number and estimate of the proportion of HCV RNA positive individuals who start treatment in the intervention vs control group
To assess the acceptability and feasibility of HCV self-testing at baseline and after study participation as assessed by responses to the questionnaire at baseline and after study participation | 2 weeks to 3 months after enrollment
  Analysis of survey responses using proportions and means. The responses to the questionnaire at baseline and after study participation will be compared to assess if there are changes in acceptability of HCV self-testing
To assess the cost of HCV self-testing | entire duration of study, estimated 6 months
  Cost per test completed, cost per person diagnosed (serology, RNA) in the intervention vs control groups. The costs of each step on the testing pathway will be combined to determine the overall cost per person diagnosed with HCV viremia

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Radzi Abu Hassan, Principal Investigator — Hospital Sultanah Bahiyah
Locations (1):
- Jom test platform, Nationally, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shilton S, Sem X, Chan HK, Chung HY, Karunanithy A, Markby J, Chan PL, Luhmann N, Johnson C, Nabeta P, Nasir NHB, Ongarello S, Reipold EI, Hassan MRA. A quasi-randomised controlled trial of online distribution of home-based hepatitis C self-testing for key populations in Malaysia: a study protocol. Trials. 2022 Apr 12;23(1):304. doi: 10.1186/s13063-022-06230-y. PMID 35413933